CLINICAL TRIAL: NCT07191548
Title: Treatment of LIVER METastases From Colorectal Cancer by IRreversible Electroporation: A Prospective, International, Multi-centre Cohort Study.
Brief Title: International Study on Treatment of Patients With Metastatic Colorectal Liver Lesions Patients With IRE
Acronym: LIVERMET-IRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ONC-01
Record Dates: First submitted 2025-09-23; First posted 2025-09-25 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Adenocarcinoma Metastatic in the Liver; Liver Ablation; Liver Cancer, Adult
Keywords: irreversible electroporation; liver ablation; metastatic liver disease; nanoknife; liver ire registry
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases | interventions — Electroporation

STUDY DESIGN:
Intervention Model Description: This is an international, prospective, multi-centre, registry-based, non-randomized, single arm, clinical cohort study of the use of IRE for the treatment of liver metastases from colorectal cancer in patients who have received systemic chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Use of NanoKnife System for ablation of metastatic colorectal lesions (Experimental)
  Interventions: Device: Irreversible Electroporation

INTERVENTIONS:
Device: Irreversible Electroporation — Irreversible electroporation (IRE) is a procedure which involves the passage of short intense electrical pulses between probes to destabilize cell membranes by creating "nanopores" which leads to cell destabilisation and cell death.
  IRE can be used to selectively damage cancerous cells whilst sparing adjacent supporting connective tissue in vessels and bile ducts allowing a more targeted treatment compared to other types of ablation. IRE also avoids the heat-sink phenomenon which compromises the effectiveness of thermal ablation and possibly reduces the risks of biliary injury.
  Other Names: nanoknife

SUMMARY:
Procedural data will be recorded from patients with liver metastases from colorectal cancer who have received at least one course of systemic chemotherapy and who have been assessed by an appropriately constituted MDT (or equivalent) as appropriate to receive irreversible electroporation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over, able to provide informed consent and with histological confirmation of a diagnosis of colorectal cancer from primary tumour.
* Liver lesions demonstrating radiological characteristics (on magnetic resonance scan) of colorectal hepatic metastases without requirement for biopsy. In the setting of an intact liver, patients with up to four metastases ≤ 4cm in size are eligible for inclusion. In the setting of proposed resection plus ablation, up to two metastases ≤ 4cm in size. In the setting of recurrence after prior hepatectomy up to two metastases ≤ 4cm in size.
* Eastern Co-operative Oncology Group (ECOG) Score ≤ 2.
* Rockwood Frailty Score ≤ 3.
* Serum bilirubin < 30 µmol/L.
* Serum creatinine < 150 µmol/L.
* Up to two lung metastases (< 2cm in size permitted at enrolment).
* Prior treatment with at least one course of systemic chemotherapy (± biologic agent) mandated. Chemotherapy protocol is not specified and is at clinician discretion.
* Primary rectal tumour can remain in situ treated with radiotherapy/chemoradiotherapy according to tumour board recommendations. Primary colonic tumour can remain in situ.
* No prior hepatic tumour ablation

Exclusion Criteria:

* Patients involved in other research studies.
* Inability to give informed consent.
* Patients who are pregnant.
* Accepted exclusions to IRE from consensus criteria including:
* Platelet count < 50x109 U/L.
* International normalised ratio (INR) for blood clotting > 1.7.
* Prior hepatic tumour ablation.

Cardiovascular fitness related exclusions:

* History of ventricular arrhythmia.
* Implanted pacemaker or defibrillator.
* Congestive cardiac failure NYHA Class ≥ 3.

Tumour-related exclusions:

* Tumour ≥ 4 cm in size.
* Advanced multi-site metastatic cancer (any of the following): peritoneal metastases (M1c), bone metastases, > 2 lung metastases, all segment involvement multiple liver metastases.
* Jaundice (serum bilirubin > 30 µmol/L).
* MDT/tumour recommends use of thermal ablation instead of IRE for any given lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Target Tumour Eradication | 6 months
  The percentage of target tumours successfully eradicated 6 months after the initial IRE procedure, according to RECIST and PERCIST criteria.

SECONDARY OUTCOMES:
Complications of IRE: Episode-related complications: | 30 days
  All complications recorded during inpatient stay recorded using Clavien-Dindo and CCI
Complications of IRE: Intervention for local liver-related complications of IRE | 12 months
  Intervention for local liver-related complications of IRE within 12 months of the procedure categorised as radiological, surgical or medical
Oncological outcomes: Local progression at site of IRE-treated lesion | 12 months
  Local progression at site of IRE-treated lesion
Oncological Outcomes: Re-ablation and modality. | 12 months
  Re-ablation and modality.
Oncological Outcomes: New lesions | 12 months
  Appearance of new lesions in liver, lungs, peritoneum or elsewhere (other) on follow-up.
Oncological Outcomes: Post IRE Chemotherapy | 12 months
  Any use of chemotherapy after IRE
Oncological Outcomes: Other liver-directed interventions | 12 months
  Any further liver-directed, anti-cancer intervention including surgery and radiotherapy.
Oncological Outcomes: Disease-free and overall survival from time of IRE. | 12 months
  Disease-free and overall survival from time of IRE.
Quality of life - pre procedure | pre procedure up to 7 days
  EQ-5D-5L survey
Quality of life - 7 days follow-up | 7 days
  EQ-5D-5L survey
Quality of life - 6 months | 6 months
  EQ-5D-5L survey

CONTACTS AND LOCATIONS:
Overall Officials: Ajith Siriwardena, MD FRCS, Principal Investigator — Manchester Royal Infirmiary
Locations (1):
- Manchester Royal Infirmiary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided